CLINICAL TRIAL: NCT02224235
Title: COBRA PZF™ Coronary Stent System in Native Coronary Arteries for Early Healing, Thrombus Inhibition, Endothelialization and Avoiding Long-term Dual Anti-platelet Therapy: OCT (Optical Coherence Tomography) Evaluation in Comparison With DES
Brief Title: COBRA SHIELD OCT Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: CeloNova BioSciences, Inc. (Industry)
Collaborators: ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COBRA 2013-02
Record Dates: First submitted 2014-08-19; First posted 2014-08-25 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Stable Angina
Keywords: Stable angina; PCI; Percutaneous Coronary Intervention
MeSH Terms: conditions — Angina, Stable | interventions — Aspirin; Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1- COBRA 1 week DAPT (Experimental): COBRA PzF coronary stent followed by dual anti-platelet therapy (DAPT) for one week
  Interventions: Device: COBRA PzF; Drug: DAPT
- Group 2 - DES 6 month DAPT (Active Comparator): Resolute Integrity DES followed by dual anti-platelet therapy (DAPT) for at least 6 months
  Interventions: Device: Resolute Integrity DES; Drug: DAPT
- Group 3 - COBRA Aspirin (Experimental): COBRA PzF coronary stent followed by aspirin alone
  Interventions: Drug: Aspirin; Device: COBRA PzF

INTERVENTIONS:
Drug: Aspirin — 75-325 mg q.d. aspirin until study completion (recommended indefinitely for stent patients)
  Other Names: Ascriptin Enteric; Aspir 81; Aspir-Low; Bufferin; Easprin; Ecotrin; Ecpirin; Fasprin; Halfprin; Miniprin
  Arms: Group 3 - COBRA Aspirin
Device: Resolute Integrity DES — Resolute Integrity DES
  Arms: Group 2 - DES 6 month DAPT
Device: COBRA PzF
  Other Names: COBRA PzF coronary stent system
  Arms: Group 1- COBRA 1 week DAPT; Group 3 - COBRA Aspirin
Drug: DAPT — At the discretion of the investigator as to which DAPT is administered (per local practice)
  Other Names: Dual Anti Platelet Therapy
  Arms: Group 1- COBRA 1 week DAPT; Group 2 - DES 6 month DAPT

SUMMARY:
Phase one of this study is a prospective, randomized (2:1), pilot study that will evaluate COBRA PzF vascular healing patterns and thrombus formation with Optical Coherence Tomography (OCT) at 3 months after stent implantation in comparison with Resolute Integrity drug eluting stent (DES). Patients in the COBRA PzF (Group 1) will receive dual anti platelets for one week followed by aspirin, while patients implanted with ZES (Group 2), will receive Dual anti-platelet therapy (DAPT) for at least 6 months followed by aspirin.

After the completion of Phase 1, Phase 2 will enroll 10 patients in the COBRA PzF (Group 3). Patients in Group 3 will receive aspirin alone and have OCT at one month after the stent procedure to evaluate COBRA PzF vascular healing patterns and thrombus formation at one month follow up.

DETAILED DESCRIPTION:
Phase one of this study is a prospective, randomized (2:1), pilot study that will evaluate COBRA PzF vascular healing patterns and thrombus formation with Optical Coherence Tomography (OCT) at 3 months after stent implantation in comparison with Resolute Integrity drug eluting stent (DES). Patients in the COBRA PzF (Group 1) will receive dual anti platelets for one week followed by aspirin, while patients implanted with ZES (Group 2), will receive Dual anti-platelet therapy (DAPT) for at least 6 months followed by aspirin.

After the completion of Phase 1, Phase 2 will enroll 10 patients in the COBRA PzF (Group 3). Patients in Group 3 will receive aspirin alone and have OCT at one month after the stent procedure to evaluate COBRA PzF vascular healing patterns and thrombus formation at one month follow up.

This study was terminated after enrollment of 8 patients due to insufficient enrollment

ELIGIBILITY:
Inclusion Criteria:

* Patient >= 18 years old.
* Eligible for percutaneous coronary intervention (PCI).
* Patient provides written informed consent.
* Patient is willing to comply with follow-up evaluation.
* Acceptable candidate for coronary artery bypass graft (CABG) surgery.
* Stable angina pectoris or a positive functional ischemia study.
* Male or non-pregnant female patient
* Patient indicated for elective stenting of up to 2 stenotic lesions in two separate native coronary arteries.
* Reference vessel >=2.5 mm and<= 4.0 mm in diameter by visual estimate.
* Target lesion <=20 mm in length by visual estimate.
* Protected left main lesion with >50% stenosis.
* Target lesion stenosis >= 70% and < 100% by visual estimate OR Target lesion stenosis <70% who meet physiological criteria for revascularization (i.e. positive Fractional Flow Reserve).

Exclusion Criteria:

* Currently enrolled in another investigational device or drug trial.
* Previously enrolled in another stent trial within the prior 2 years.
* ANY planned elective surgery or percutaneous intervention within the subsequent 3 months.
* A previous coronary interventional procedure of any kind within 30 days prior to the procedure.
* The patient requires staged procedure of either the target or any non-target vessel before OCT procedure at 3 months post-procedure.
* The target lesion requires treatment with a device other than percutaneous transluminal coronary angioplasty (PTCA) prior to stent placement.
* Previous drug eluting stent (DES) or bare metal stent (BMS) deployment anywhere in the target vessel.
* Co-morbid condition(s) that could limit the patient's ability to participate in the trial or to comply with follow-up requirements, or impact the scientific integrity of the trial.
* Concurrent medical condition with a life expectancy of less than 12 months.
* Documented left ventricular ejection fraction (LVEF) < 50% at the most recent evaluation.
* Patients with diagnosis of myocardial infarction (MI) within 72 hours (i.e. CK-MB must be returned to normal prior to enrollment) or suspected acute MI at time of enrollment.
* Previous intervention in the target vessel.
* History of cerebrovascular accident or transient ischemic attack in the last 6 months.
* Leukopenia (leukocytes < 3.5 x10^9 / liter).
* Neutropenia (Absolute Neutrophil Count < 1000/mm3) <= 3 days prior to enrollment.
* Thrombocytopenia (platelets < 100,000/mm3) pre-procedure.
* Active peptic ulcer or active GI bleeding.
* History of bleeding diathesis or coagulopathy or inability to accept blood transfusions.
* Known hypersensitivity or contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, L-605 Cobalt chromium alloy or sensitivity to contrast media, which cannot be adequately pre-medicated.
* Serum creatinine level > 2.0 mg/dl within 7 days prior to index procedure.
* Patients not responsive to Plavix/ aspirin and or unable to tolerate Plavix/ aspirin for 6 month post procedure.
* Patient on or may require anticoagulation therapy within 3 months of index procedure.
* Flow limiting dissections observed on OCT
* Significant tissue prolapse within the stent observed on OCT
* Unprotected left main coronary artery disease
* Target vessel with any lesions with greater than 60% diameter stenosis outside of a range of 5 mm proximal and distal to the target lesion based on visual estimate or on-line quantitative coronary arteriography (QCA).
* Target lesion (or vessel) exhibiting an intraluminal thrombus (occupying > 50% of the true lumen diameter) at any time.
* Lesion location that is aorto-ostial or within 5 mm of the origin of the left anterior descending (LAD) or left circumflex (LCX).
* Target lesion with side branches > 2.0mm in diameter.
* Target vessel is excessively tortuous (two bends > 90˚ to reach the target lesion).
* Target lesion is severely calcified.
* Thrombolysis In Myocardial Infarction (TIMI) flow 0 or 1
* Target lesion is in a bypass graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neointimal coverage of the stent as measured using OCT | 1 month
  Neointimal coverage of the stent as measured using OCT
Neointimal coverage of the stent as measured using OCT | 3 months
  Neointimal coverage of the stent as measured using OCT
Presence of thrombus formation as measured by OCT | 1 month
  Presence of thrombus formation as measured by OCT
Presence of thrombus formation as measured by OCT | 3 months
  Presence of thrombus formation as measured by OCT
Proportion of uncovered struts as measured by OCT | 1 month
  Proportion of uncovered struts as measured by OCT
Proportion of uncovered struts as measured by OCT | 3 months
  Proportion of uncovered struts as measured by OCT
Presence of Malopposed struts as measured by OCT | 1 month
  Presence of Malopposed struts as measured by OCT
Presence of Malopposed struts as measured by OCT | 3 months
  Presence of Malopposed struts as measured by OCT
In-stent neointimal thickness measured using OCT | 1 month
  In-stent neointimal thickness measured using OCT
In-stent neointimal thickness measured by OCT | 3 months
  In-stent neointimal thickness measured by OCT
Lumen area measured by OCT | 1 month
  Lumen area measured by OCT
Lumen area measured by OCT | 3 months
  Lumen area measured by OCT
Lumen Volume measured by OCT | 1 month
  Lumen Volume measured by OCT
Lumen Volume measured by OCT | 3 months
  Lumen Volume measured by OCT
Stent area measured by OCT | 1 month
  Stent area measured by OCT
Stent area measured by OCT | 3 months
  Stent area measured by OCT
Stent volume measured by OCT | 1 month
  Stent volume measured by OCT
Stent volume measured by OCT | 3 months
  Stent volume measured by OCT

OTHER OUTCOMES:
In-stent late loss measured by angiography | 1 month
  In-stent late loss measured by angiography
In-stent late loss measured by angiography | 3 months
  In-stent late loss measured by angiography
In-segment late loss measured by angiography | 1 month
  In-segment late loss measured by angiography
In-segment late loss measured by angiography | 3 months
  In-segment late loss measured by angiography
In-stent percent diameter stenosis measured by angiography | 1 month
  In-stent percent diameter stenosis (%DS) measured by angiography
In-stent percent diameter stenosis measured by angiography | 3 months
  In-stent percent diameter stenosis (%DS) measured by angiography
In-segment percent diameter stenosis measured by angiography | 1 month
  In-segment percent diameter stenosis measured by angiography (%DS) (within the 5 mm margins proximal and distal to stent)
In-segment percent diameter stenosis measured by angiography | 3 months
  In-segment percent diameter stenosis measured by angiography (%DS) (within the 5 mm margins proximal and distal to stent)
In-stent binary stenosis measured by angiography | 1 month
  In-stent binary stenosis measured by angiography
In-stent binary stenosis measured by angiography | 3 months
  In-stent binary stenosis measured by angiography(stenosis of > 50% of the reference vessel diameter)
In-segment binary stenosis measured by angiography | 1 month
  In-segment binary stenosis measured by angiography (stenosis of > 50% of the reference vessel diameter)
In-segment binary stenosis measured by angiography | 3 months
  In-segment binary stenosis measured by angiography (stenosis of > 50% of the reference vessel diameter)
In-stent minimum lumen diameter measured by angiography | 1 month
  In-stent minimum lumen diameter (MLD) measured by angiography
n-stent minimum lumen diameter measured by angiography | 3 months
  In-stent minimum lumen diameter (MLD) measured by angiography
In-segment minimum lumen diameter (MLD) measured by angiography | 1 month
  In-segment MLD measured by angiography
In-segment minimum lumen diameter (MLD) measured by angiography | 3 months
  In-segment MLD measured by angiography
Longitudinal stent deformation measured by angiography | 1 month
  Longitudinal stent deformation measured by angiography
Longitudinal stent deformation measured by angiography | 3 months
  Longitudinal stent deformation measured by angiography
Presence of stent fracture measured by angiography | 1 month
  Presence of stent fracture measured by angiography
Presence of stent fracture measured by angiography | 3 months
  Presence of stent fracture measured by angiography
All Deaths | 1 month
  All Deaths from any cause post index procedure
All Deaths | 6 months
  All Deaths from any cause post index procedure
All Deaths | 12 months
  All Deaths from any cause post index procedure
Cardiac Death | 1 month
  Death due to cardiac cause post index procedure
Cardiac Death | 6 months
  Death due to cardiac cause post index procedure
Cardiac Death | 12 months
  Death due to cardiac cause post index procedure
Major Adverse Cardiac Events | 1 month
  Major Adverse Cardiac Events (MACE) defined as cardiac death, MI (Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods
Major Adverse Cardiac Events | 6 months
  Major Adverse Cardiac Events (MACE) defined as cardiac death, MI (Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods
Major Adverse Cardiac Events | 12 months
  Major Adverse Cardiac Events (MACE) defined as cardiac death, MI (Q wave and non-Q wave), emergent bypass surgery, or clinically driven target lesion revascularization (TLR) by percutaneous or surgical methods
Myocardial Infarction | 1 month
  Occurrence of myocardial infarction. Defined as either a Q wave MI (QWMI) or Non-Q wave MI (NQWMI).
Myocardial Infarction | 6 months
  Occurrence of myocardial infarction. Defined as either a Q wave MI (QWMI) or Non-Q wave MI (NQWMI).
Myocardial Infarction | 12 months
  Occurrence of myocardial infarction. Defined as either a Q wave MI (QWMI) or Non-Q wave MI (NQWMI).
Composite endpoint of cardiac death and MI | 1 month
  Composite endpoint of Cardiac Death and MI
Composite endpoint of cardiac death and MI | 6 months
  Composite endpoint of Cardiac Death and MI
Composite endpoint of cardiac death and MI | 12 months
  Composite endpoint of Cardiac Death and MI
Clinically driven Target Lesion Revascularization | 1 month
  Clinically driven TLR. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Clinically driven Target Lesion Revascularization | 6 months
  Clinically driven TLR. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Clinically driven Target Lesion Revascularization | 12 months
  Clinically driven TLR. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the stent.
Clinically driven target vessel revascularization | 1 month
  Clinically driven TVR. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
Clinically driven target vessel revascularization | 6 months
  Clinically driven TVR. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
Clinically driven target vessel revascularization | 12 months
  Clinically driven TVR. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches and the target lesion itself.
Occurrence of Stroke post index procedure | 1 month
  Stroke (ischemic and hemorrhagic)
Occurrence of Stroke post index procedure | 6 months
  Stroke (ischemic and hemorrhagic)
Occurrence of Stroke post index procedure | 12 months
  Stroke (ischemic and hemorrhagic)
Acute success | 30 days
  Device Success: Defined as the attainment of < 30% final residual stenosis of the target lesion using only the COBRA PzFTM Coronary Stent System Lesion Success: Defined as the attainment of < 30% final residual stenosis of the target lesion using any percutaneous method.
  Procedure Success: Attainment of < 30% residual stenosis of the target lesion and no in-hospital MACE.
Bleeding or vascular complications | At time of hospital discharge (expected average to be within 2 days of index procedure
  Bleeding Complications: Defined as a procedure-related hemorrhagic event that requires a transfusion and/or surgical intervention.
  Vascular Complications may include pseudoaneurysm, arteriovenous fistula (AVF), peripheral ischemia/nerve injury, and vascular event requiring transfusion or surgical repair.
Stent Thrombosis | 3 months
  Stent Thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the patient has left the catheterization laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi Karjalainen, MD, PhD, Principal Investigator — Satakunta Central Hospital
Locations (2):
- Finland (2):
  - Satakunta Central Hospital, Pori
  - Heart Center, Turku University Hospital, Turku